CLINICAL TRIAL: NCT06369727
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of MOB015B in Healthy Subjects Using a Repeat Insult Patch Test Design
Brief Title: Study to Evaluate the Sensitizing Potential of MOB015B in Healthy Subjects Using a Repeat Insult Patch Test Design
Acronym: RIPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MOB015B-VI
Record Dates: First submitted 2017-08-01; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Erythema
MeSH Terms: conditions — Erythema | interventions — Sodium Chloride

STUDY DESIGN:
Masking Description: NA- Safety study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MOB015B (Experimental): Patches were applied to the infrascapular area
  Interventions: Drug: MOB015B
- Vehicle (Placebo Comparator): Patches were applied to the infrascapular area
  Interventions: Drug: MOB015B vehicle
- Negative irritant solution (0.9% saline) (Other): Patches were applied to the infrascapular area
  Interventions: Drug: Negative irritant solution of 0.9% saline

INTERVENTIONS:
Drug: MOB015B — Topcal formulation
  Arms: MOB015B
Drug: MOB015B vehicle — Topcal formulation
  Arms: Vehicle
Drug: Negative irritant solution of 0.9% saline — Negative control
  Arms: Negative irritant solution (0.9% saline)

SUMMARY:
A Randomized, Controlled Study to Evaluate the Sensitizing Potential of MOB015B in Healthy Subjects Using a Repeat Insult Patch Test Design To evaluate the sensitization potential

DETAILED DESCRIPTION:
MOB015B is a topical solution for the treatment of nail fungus (onychomycosis) containing the active antifungal ingredient terbinafine. Terbinafine is a well-known antifungal agent that has been widely used for decades for both in topical and oral preparations and is regarded as an effective treatment of dermatophyte infections. In a phase II study, MOB015B was found to be efficacious and safe in the topical treatment of distal subungual onychomycosis. This Phase 1 study will assess the sensitization potential of MOB015B.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female (to be confirmed by medical history);
2. Is 18 years of age or older;
3. In the case of a female of childbearing potential, is using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy, tubal ligation). Abstinence or vasectomies are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
4. In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) on Day 1 prior to randomization and are willing to submit to a UPT at the end of study (EOS);
5. Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs;
6. Is of any Fitzpatrick Skin Type or race, providing the skin pigmentation will allow discernment of erythema (see Table 1);
7. Complete a medical screening procedure; and
8. Read, understand, and sign an informed consent.

Exclusion Criteria:

1. Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction;
2. Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
3. Is not willing to refrain from using systemic/topical anti-inflammatory analgesics such as aspirin (81 mg daily aspirin will be allowed), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
4. Is using medication which, in the opinion of the Investigator, will interfere with the study results (e.g. anti-inflammatory medications, antipsychotics, anticonvulsants with potential pain relief effects, immunomodulatory medications, and others);
5. Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study;
6. Has psoriasis and/or active atopic dermatitis/eczema;
7. Has a known sensitivity or allergy to constituents of the materials being evaluated;
8. Is a female who is pregnant, plan to become pregnant during the study, or is breast feeding a child;
9. Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
10. Has received treatment for any type of internal cancer within 5 years prior to study entry;
11. Has a history of, or are currently being treated for skin cancer and/or hepatitis;
12. Has a history of, or is currently being treated for, insulin dependent diabetes;
13. Has any condition that might compromise study results;
14. Currently or expect to sunbathe or use tanning salons during the study;
15. Is currently participating in any clinical testing;
16. Has any known sensitivity to adhesives; and/or
17. Has received any investigational drug(s) within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
To determine the potential of MOB015B to induce sensitization by repeated topical application to the healthy skin of humans under controlled conditions. | 6 weeks
  Evaluation of dermal reactions at the application sites assessed clinically using a visual scale that rates the degree of erythema, edema, and other signs of cutaneous irritation.
To assess safety | 6 weeks
  Evaluation of any adverse events (AEs) reported during the study.application to the healthy skin of humans.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Inc, Fair Lawn, New Jersey, United States